CLINICAL TRIAL: NCT05691998
Title: Comparison of Different Types of Prosthetic Foot: Patient Perspective
Brief Title: Comparison of Different Types of Prosthetic Foott
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associated Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 33
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: the Previous Prosthetic Foot Experience of Patients With Amputation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: the previous prosthesis experience
  Interventions: Other: Prosthetic foot questionnaire

INTERVENTIONS:
Other: Prosthetic foot questionnaire — Prosthetic foot related questions will be asked to the patients

SUMMARY:
The main purpose of this study is to determine the experiences of patients with different types of prostetic feet (carbon, hydraulic or microprocessor controlled).

DETAILED DESCRIPTION:
One of the main goals in the rehabilitation of amputees is to provide optimal and natural ambulation. For this purpose, suitable socket-suspension type, appropriate knee joint and foot should be prescribed. In the selection of feet, the age, occupation, characteristics of the geographical region, mental status and activity level should be considered. In addition, the previous prosthesis experience of the people should definitely be taken into account during prosthesis prescribing.The main purpose of this study is to determine the experiences of patients with different types of prostetic feet (carbon, hydraulic or microprocessor controlled).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years
* Lower limb amputation
* Having used at least 2 different foot types (carbon, hydrolic, microprocessor-controlled)

Exclusion Criteria:

* Having used the single type of foot until now
* Presence of neurological, cardiovascular, and pulmonary disease that may affect walking performance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 patients with lower limb amputation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-01-25 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Qestion 1 | through study completion, an average of one and a half months
  Walking on the straight road
Qestion 2 | through study completion, an average of one and a half months
  Walking on uneven terrain

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Demir, Associated Professor, Principal Investigator — dr_yasindemir@yahoo.com

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilinc Kamaci G, Artuc SE, Ceylan H, Tekin E, Kanlioglu O, Orucu Atar M, Demir Y, Aydemir K. Comparison of different types of prosthetic feet in patients with unilateral transtibial amputation; patient perspective. J Orthop Sci. 2025 Aug 13:S0949-2658(25)00207-6. doi: 10.1016/j.jos.2025.07.007. Online ahead of print. PMID 40813189